CLINICAL TRIAL: NCT01232465
Title: Impact of Sperm DNA Integrity on In Vitro Cycles
Acronym: TBA on IVF
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 10-249A
Record Dates: First submitted 2010-10-28; First posted 2010-11-02 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-03

CONDITIONS: Male Infertility; Unexplained Infertility; Abortion, Habitual
Keywords: sperm DNA integrity; Toluidine blue assay (TBA); IVF outcome
MeSH Terms: conditions — Infertility, Male; Abortion, Habitual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — slide smears will be kept to observe overall DNA integrity of sperm sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IVF: those individuals undergoing conventional IVF to inseminate their retrieved eggs
- ICSI: those individuals whose eggs were fertilized via intracytoplasmic sperm injection (ICSI)

SUMMARY:
Sperm DNA integrity will be measured via the Toluidine Blue Assay (TBA) for patients undergoing In Vitro Fertilization (IVF); the study will determine correlations, if any, between IVF success and sperm DNA integrity.

ELIGIBILITY:
Inclusion Criteria:

* couple undergoing IVF at the Center for Human Reproduction
* sperm sample given from partner (not a donor)

Exclusion Criteria:

* low sperm concentration (<5 million/cc)
* using a donor sample

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: couples undergoing IVF treatement at the Center for Human Reproduction, North Shore University Hospital, Manhasset NY
Sampling Method: Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avner E Hershlag, MD, Principal Investigator — Center for Human Reproduction
Locations (1):
- Center for Human Reproduction, Manhasset, New York, United States

REFERENCES:
- [Background] Andreetta AM, Stockert JC, Barrera C. A simple method to detect sperm chromatin abnormalities: cytochemical mechanism and possible value in predicting semen quality in assisted reproductive procedures. Int J Androl. 1995 Jun;18 Suppl 1:23-8. doi: 10.1111/j.1365-2605.1995.tb00634.x. PMID 7558384
- [Background] Erenpreisa J, Erenpreiss J, Freivalds T, Slaidina M, Krampe R, Butikova J, Ivanov A, Pjanova D. Toluidine blue test for sperm DNA integrity and elaboration of image cytometry algorithm. Cytometry A. 2003 Mar;52(1):19-27. doi: 10.1002/cyto.a.10015. PMID 12596248
- [Background] Erenpreiss J, Bars J, Lipatnikova V, Erenpreisa J, Zalkalns J. Comparative study of cytochemical tests for sperm chromatin integrity. J Androl. 2001 Jan-Feb;22(1):45-53. PMID 11191087
- [Background] Erenpreiss J, Jepson K, Giwercman A, Tsarev I, Erenpreisa J, Spano M. Toluidine blue cytometry test for sperm DNA conformation: comparison with the flow cytometric sperm chromatin structure and TUNEL assays. Hum Reprod. 2004 Oct;19(10):2277-82. doi: 10.1093/humrep/deh417. Epub 2004 Jul 22. PMID 15271869
- [Background] Schlegel PN, Paduch DA. Yet another test of sperm chromatin structure. Fertil Steril. 2005 Oct;84(4):854-9. doi: 10.1016/j.fertnstert.2005.04.050. PMID 16213834
- [Background] Collins JA, Barnhart KT, Schlegel PN. Do sperm DNA integrity tests predict pregnancy with in vitro fertilization? Fertil Steril. 2008 Apr;89(4):823-31. doi: 10.1016/j.fertnstert.2007.04.055. Epub 2007 Jul 20. PMID 17644094
- [Background] Simon L, Brunborg G, Stevenson M, Lutton D, McManus J, Lewis SE. Clinical significance of sperm DNA damage in assisted reproduction outcome. Hum Reprod. 2010 Jul;25(7):1594-608. doi: 10.1093/humrep/deq103. Epub 2010 May 6. PMID 20447937
- [Background] Tarozzi N, Bizzaro D, Flamigni C, Borini A. Clinical relevance of sperm DNA damage in assisted reproduction. Reprod Biomed Online. 2007 Jun;14(6):746-57. doi: 10.1016/s1472-6483(10)60678-5. PMID 17579991
- [Background] Zini A, Libman J. Sperm DNA damage: clinical significance in the era of assisted reproduction. CMAJ. 2006 Aug 29;175(5):495-500. doi: 10.1503/cmaj.060218. PMID 16940270
- [Background] Sharma RK, Said T, Agarwal A. Sperm DNA damage and its clinical relevance in assessing reproductive outcome. Asian J Androl. 2004 Jun;6(2):139-48. PMID 15154089
- [Background] Speyer BE, Pizzey AR, Ranieri M, Joshi R, Delhanty JD, Serhal P. Fall in implantation rates following ICSI with sperm with high DNA fragmentation. Hum Reprod. 2010 Jul;25(7):1609-18. doi: 10.1093/humrep/deq116. Epub 2010 May 22. PMID 20495207
- [Background] Tsarev I, Bungum M, Giwercman A, Erenpreisa J, Ebessen T, Ernst E, Erenpreiss J. Evaluation of male fertility potential by Toluidine Blue test for sperm chromatin structure assessment. Hum Reprod. 2009 Jul;24(7):1569-74. doi: 10.1093/humrep/dep068. Epub 2009 Mar 21. PMID 19304993

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occured at the Center for Human Reproduction under an IRB waiver of informed consent for participation.
Groups:
- IVF Cycles: those individuals undergoing conventional IVF to inseminate their retrieved eggs
Period: Overall Study
Arm/Group | IVF Cycles | ICSI
Started | 337 | 402
Completed | 337 | 402
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVF Cycles | ICSI | Total
Number analyzed (Participants) | 337 | 402 | 739
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 337 | 402 | 739
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (2.6) | 34.9 (2.5) | 34.8 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 337 | 402 | 739
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 337 | 402 | 739

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy
Description: detemining whether the sperm sample (tested for DNA integrity) used to insemenate IVF retrieved eggs, results in a live birth
Time Frame: 9 months
Measure: Number; unit: participants
Arm/Group | IVF Cycles | ICSI
Number analyzed (Participants) | 337 | 402
participants | 67 | 80

ADVERSE EVENTS:
Description: Measurements of sperm DNA integrity did not have an impact on cycle treatment, failure or success. There were no adverse events in obtaining this data, as the samples were already submitted for clinical purposes. A small aliquat was removed from the clinical sample to generate study data.
Arm/Group | IVF Cycles | ICSI
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes